CLINICAL TRIAL: NCT01387243
Title: Survey on the Pharmacy Follow up of Alli Purchasers
Brief Title: Survey on the Pharmacy Follow-up of Alli Purchasers
Status: Completed | Type: Observational
Sponsor: GlaxoSmithKline (Industry)
Responsible Party: Sponsor
Other Study IDs: W5350856
Record Dates: First submitted 2010-03-29; First posted 2011-07-04 (Estimated); Last update posted 2012-10-29 (Estimated); Status verified 2012-10

CONDITIONS: Overweight
Keywords: behavior modification; overweight; orlistat
MeSH Terms: conditions — Overweight | interventions — Orlistat

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- 60 mg Orlistat: Purchased by consumer
  Interventions: Drug: Orlistat

INTERVENTIONS:
Drug: Orlistat — 60 mg

SUMMARY:
To assess the feasibility and acceptability of genuine pharmacy follow up of people wishing to lose weight.

ELIGIBILITY:
Inclusion Criteria:

* Individuals who have been recognized as being eligible for treatment, who have agreed to pharmacy follow up, and have given their informed consent to take part in the survey.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Consumers purchasing orlistat in a pharmacy setting
Sampling Method: Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2010-01; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
Change in Physical activity | baseline to 1 year

SECONDARY OUTCOMES:
Change in dietary behavior | baseline to 1 year
Evaluation of care pathway (e.g., consultation with doctors, use of nutritional information) | baseline to 1 year
Satisfaction with management (i.e., results on weight and treatment comfort) | baseline to 1 year

CONTACTS AND LOCATIONS:
Overall Officials: GSK Clinical Trials, Study Director — GlaxoSmithKline